CLINICAL TRIAL: NCT00501748
Title: Open Label Study of Safety and Tolerability of Rituximab in Neuromyelitis Optica, Recurrent Transverse Myelitis and Recurrent Bilateral Simultaneous Optic Neuritis
Brief Title: Safety and Tolerability of Rituximab in Neuromyelitis Optica
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H7620-25392-04
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Neuromyelitis Optica
Keywords: Neuromyelitis Optica; acute transverse myelitis
MeSH Terms: conditions — Neuromyelitis Optica; Myelitis, Transverse | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab is a highly purified, 1328-amino acid antibody with an approximate molecular mass of 145 kD. Rituximab is a sterile, clear, colorless, preservative-free liquid concentrate for intravenous (IV) administration. Rituximab is supplied at a concentration of 10 mg/mL in either 100 mg (10 mL) or 500 mg (50 mL) single-use vials. In this single arm study all subjects are treated with two cycles of rituximab. Each cycle consists of two 1000 mg infusions administered two weeks apart. The cycles of rituximab treatment are administered at baseline and at 9 months.
  Other Names: Rituxan

SUMMARY:
The goal of this research study is to investigate whether Rituximab is safe to use in patients suffering from NMO, or who are at high risk for developing NMO. It is thought that NMO is caused by the immune system reacting against the optic nerves and spinal cord. B cells are a part of the immune system that may contribute to the illness. Rituximab is an antibody that depletes B cells. Depletion of these B cells with Rituximab may induce remission of the disease. Because pathological and serological studies suggest that NMO appears to be, at least in part, a B-cell mediated disease Rituximab, is an attractive treatment candidate for this disease.

DETAILED DESCRIPTION:
Rituximab is a genetically engineered, chimeric, murine/human monoclonal antibody directed against the CD20 antigen found on the surface of normal and malignant pre-B and mature B cells. The antibody is an IgG1 immunoglobulin containing murine light- and heavy chain variable region sequences and human constant region sequences. Rituximab is composed of two heavy chains of 451 amino acids and two light chains of 213 amino acids (based on cDNA analysis) and has an approximate molecular mass of 145 kD. Rituximab has a binding affinity for the CD20 antigen of ~8.0 nM.

Rituximab was developed by Biogen Idec and Genentech, Inc. It was approved by the FDA in 1997 for the treatment of relapsed or refractory low grade or follicular, CD20+, B-cell non-Hodgkin's lymphoma (NHL).

Rituximab has also been studied in a variety of non-malignant autoimmune disorders where B cells and auto antibodies appear to play a role in pathophysiology. Rituximab has been reported to relieve signs and symptoms of rheumatoid arthritis , lupus , immune thrombocytopenia , autoimmune anemia , autoimmune neuropathy , and paraneoplastic opsoclonus/myoclonus .

A Phase II study (WA16291) has been completed in patients with rheumatoid arthritis (RA) . A total of 161 patients were randomized to 4 treatment arms: Methotrexate, Rituximab alone, Rituximab and Methotrexate, Rituximab and Cyclophosphamide. Two doses of Rituximab, 1 gm each, were administered IV two weeks apart. Infusion reactions were observed in 36% of patients during their first infusion of Rituximab compared to 30% for placebo . Four Rituximab-treated patients developed serious infections, for a rate of 4.6 per 100 patient years. For context, the rate of infections requiring hospital admission was 9.57 per 100 patient years in a community based epidemiologic study in RA.

We treated 8 patients with NMO with Rituximab and observed that Rituximab appears to be well tolerated with 0/8 of the patients suffering serious adverse reactions that could be directly related to Rituximab administration. Moreover, 7/8 patients experienced decrease in neurological disability following treatment, suggesting that B-cell depletion may enhance neurological recovery from attacks. 7/8 of the patients remained attack-free within a period of 18 months of follow-up on average (range 3 to 12 months) following treatment. We observed one attack following treatment in a single patient, whereas 14 attacks would have been predicted by the pre-treatment attack rate (p=0.012, paired t test comparing pre- and post-treatment attack rates). Nevertheless, the observed impact of treatment on recovery is more than what would be expected from spontaneous recovery and deserves further investigation. If B cells are essential for pathogenesis of recurrent attacks in NMO, B cell depletion may induce sustained remission. We also observed in one case, a dramatic recovery of electrophysiological conduction in the optic nerves (visual evoked potentials), which implies that in this case, rituxan did not impair repair mechanisms, for example, demyelination following the acute attack.

ELIGIBILITY:
Inclusion criteria

1. Criteria for neuromyelitis optica:

   1. acute transverse myelitis and optic neuritis occurring within 30 days of each other followed by a second attack of either optic neuritis and/or acute transverse myelitis at least 3 months following the heralding attack OR
   2. acute transverse myelitis followed by optic neuritis at least 3 months later OR
   3. optic neuritis followed by acute transverse myelitis at least 3 months later
2. Criteria for high risk for neuromyelitis optica:

   1. recurrent idiopathic recurrent acute transverse myelitis with at least 3 months time between each attack OR
   2. recurrent bilateral simultaneous optic neuritis with at least 3 months time between each attack.

      * Subjects should also have no clinical evidence of disease outside the optic nerve or spinal cord.
      * In addition patients should have one major supportive criteria OR two minor supportive criteria:

        1. Negative brain MRI at onset (Does not meet criteria for multiple sclerosis (Paty, 1998)
        2. Spinal cord MRI with signal abnormality extending over ≥3 vertebral segments
        3. CSF pleocytosis of > 50 WBC/mm3 OR > 5 PMNs/mm3
      * Minor supportive criteria:

        1. Bilateral optic neuritis
        2. Severe optic neuritis with fixed visual acuity worse than 20/200 in at least one eye
        3. Severe, fixed, attack-related weakness (MRC ≤2) in one or more limbs
      * Subjects must have exhibited evidence of treatment failure, defined as at least one attack of either acute transverse myelitis or optic neuritis within six months of screening despite treatment within steroids or other immunomodulatory drug for the preceding attack.
      * Able and willing to give written informed consent and comply with the requirements of the study protocol.
      * Adequate renal function as indicated by normal serum sodium, potassium, chloride, bicarbonate, creatinine, and blood urea nitrogen studies.
      * Adequate liver function, as indicated by normal bilirubin and alkaline phosphatase, and transaminases (AST and ALT) within 2X upper limit of normal.
      * Negative serum pregnancy test (for women of child bearing age).
      * Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of treatment.

Exclusion Criteria:

1. Treatment with broad-spectrum immunosuppressant medications such as cyclophosphamide, mitoxantrone, methotrexate, azathioprine, and cladribine, within 60 days of screening.
2. Treatment with any investigational agent within 4 weeks of screening
3. Receipt of a live vaccine within 4 weeks prior to randomization
4. Previous Treatment with Rituximab (MabThera® / Rituxan®)
5. Prior antibody therapy
6. History of exposure to clioquinol
7. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
8. History of HIV (positive HIV, HIV conducted during screening if applicable)
9. History of Hepatitis B and/or Hepatitis C (Hep B/C at screening)
10. History of recurrent significant infection or history of recurrent bacterial infections
11. Known active bacterial, viral fungal mycobacterial, or other infection or any major episode of infection requiring hospitalization
12. Ongoing daily steroid use
13. History of drug, alcohol, or chemical abuse within 6 months prior to screening
14. Pregnancy (a negative serum pregnancy test should be performed for all women of childbearing potential within 7 days of treatment) or lactation
15. Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
16. History of psychiatric disorder

Ages: 12 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of Rituximab in NMO (monitor for any AE during two years of follow up) | 96 weeks

SECONDARY OUTCOMES:
Time from treatment to recurrence of either optic neuritis or myelitis | 96 weeks
Change in Kurtzke expanded disability status scale (EDSS) at weeks 4, 12, 24, 48, 72, 96 | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Cree, MD, PhD, Principal Investigator — MS Center , UCSF
Locations (2):
- United States (2):
  - UCSF MS Center , 350 Parnassus Ave , suite #908, San Francisco, California
  - The Neurological Institute of New York MS Center, Columbia University Medical Center 710 West 168th Street,, New York